CLINICAL TRIAL: NCT04194749
Title: Physical Therapy After Distal Radius Fracture; Traditional Versus Digital Media Based Therapy Protocol
Brief Title: Digital Media Based Physical Therapy Post Distal Radius Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Adam J. MIrarchi, Associate Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11330
Record Dates: First submitted 2019-12-02; First posted 2019-12-11 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Distal Radius Fracture
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Media Therapy (Experimental): The digital media based group will receive a modified post immobilization protocol. This will include giving the patients a Universal Serial Bus (USB) drive loaded with a 12 week physical therapy protocol presented in digital form with videos and graphical representations of exercises to be done. They will also have access to the videos and multimedia on the Oregon Health & Science University website.
  Interventions: Other: Digital Media Based Physical Therapy
- Traditional Therapy (Active Comparator): The traditional group will have clinic-based physical therapy protocol.
  Interventions: Other: Traditional Physical Therapy

INTERVENTIONS:
Other: Digital Media Based Physical Therapy — This intervention is a modified post immobilization protocol. This will include giving the patients a USB drive loaded with a 12 week therapy protocol presented in digital form with videos and graphical representations of exercises to be done. They will also have access to the videos and multimedia on the Oregon Health & Science University website.
  Arms: Digital Media Therapy
Other: Traditional Physical Therapy — This intervention is a 12 week therapist supervised clinic-based therapy protocol.
  Arms: Traditional Therapy

SUMMARY:
This trial aims to develop and test the efficacy of a digital media based physical therapy protocol on patients after surgical fixation and non-operative treatment of distal radius fractures.It is hypothesized that there will not be a difference in outcomes for patients after surgical fixation of distal radius fractures with traditional physical therapy and digital media based therapy

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing operative treatment for distal radius fractures.

Exclusion Criteria:

* Poly-trauma patients with significant previous diagnosis of dementia, previous traumatic brain injury, or other reason for significant altered mental status that would interfere with their participation in therapist directed or digital based therapy will be excluded.
* Patients who present to Oregon Health & Science University for physical therapy who will be treated by a physician at another non Oregon Health & Science University facility will be excluded.
* Patients who are not proficient in the English language will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Abbreviated version of the Disabilities of the Arm, Shoulder and Hand (QuickDASH) | 12 weeks
  Patient-Reported Outcome, Scale: 0 (no disability) - 100 (most severe disability)

SECONDARY OUTCOMES:
Abbreviated version of the Disabilities of the Arm, Shoulder and Hand (QuickDASH) | 6 weeks, 6 months
  Patient-Reported Outcome, Scale: 0 (no disability) - 100 (most severe disability)
Visual Analog Pain Scale | 6 weeks, 12 weeks, and 6 months
  Patient-Reported Outcome, Scale: 0 (no pain) - 10 (most severe pain)
Veterans RAND 12-item Health Survey (VR-12) | 6 weeks, 12 weeks, and 6 months
  Patient-Reported Outcome
Wrist Range of Motion | 6 weeks, 12 weeks, and 6 months
  Wrist flexion, extension, pronation, supination, ulnar deviation, radial deviation
Hand Grip Strength | 6 weeks, 12 weeks, and 6 months
  Strength measurement
Wrist Circumference | 6 weeks, 12 weeks, and 6 months
  Anthropometric measurement

IPD SHARING:
Plan to Share IPD: No